CLINICAL TRIAL: NCT03947918
Title: Sleep Duration and Risk for Obesity in Mexican American Children
Brief Title: Summertime: Kids in Motion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to challenges regarding COVID-19, it was not possible to reach the study's target sample size.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1K01HL129087-01A1 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-05-13 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Three-week study includes:
  Week 1 - all children get usual sleep Tuesday-Friday.
  Week 2 - children are randomized to getting no more than 8 hours or at least 10 hours of sleep (Tuesday-Friday).
  Week 3 - children crossover to the opposite sleep condition (Tuesday-Friday).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short sleep (Experimental): No more than 8 hours of sleep for 4 consecutive nights.
  Interventions: Behavioral: Short sleep; Behavioral: Long sleep
- Long sleep (Experimental): At least 10 hours of sleep for 4 consecutive nights
  Interventions: Behavioral: Short sleep; Behavioral: Long sleep

INTERVENTIONS:
Behavioral: Short sleep — Child will be asked to sleep for less than 8 hours. Study team will help parent design a sleep schedule for that week. Study team will send parent daily text messages or phone call reminders.
  Other Names: Restricted sleep
Behavioral: Long sleep — Child will be asked to sleep for more than 10 hours. Study team will help parent design a sleep schedule for that week. Study team will send parent text messages or phone call reminders.
  Other Names: Healthy sleep

SUMMARY:
This is a 3-week randomized crossover study to determine the effect of the prior night's sleep duration on energy-balance related behaviors of diet and physical activity the following day. In Week 1, child participants will sleep their usual amount. In week 2, participants will be randomized to either a sleep restricted or a healthy sleep condition for 4 nights. In week 3, participants will cross over to the opposite sleep condition for 4 nights.

DETAILED DESCRIPTION:
Individuals of Mexican descent comprise the largest proportion of the Latino population in the United States and they suffer high rates of obesity. Short sleep is a risk factor for obesity. An improved understanding of the underlying behavioral mechanisms by which short sleep duration may impact obesity among Mexican American children is critical to prevent and/or reduce obesity and chronic disease in this population. This research will focus on behavioral mechanisms (i.e., diet and physical activity) that link sleep duration to obesity. Mexican American 8-10-year-olds will participate in a 3-week crossover study to examine: 1) contextual factors (i.e., bedtime routines, sleep hygiene, familism) that may impact sleep; and 2) the impact of prior night's sleep duration on diet and physical activity the subsequent day. This research design will make it possible to examine whether sufficient sleep is protective of energy balance (e.g., healthful dietary intake/patterns and physical activity) as well as contextual factors related sleep.

ELIGIBILITY:
Inclusion Criteria:

* Mexican American child-mother pairs which will include: child 8-10 years old; mother/female guardian; English/Spanish speakers; mobile phone user.

Exclusion Criteria:

* Children with major illnesses and/or with sleep apnea for which children
* In families where 2 children are eligible for participation, a child will be selected at random to participate in the study.
* The investigators will exclude fathers from this study for reasons due to statistical power

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-06-17 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Martinez, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beebe DW, Simon S, Summer S, Hemmer S, Strotman D, Dolan LM. Dietary intake following experimentally restricted sleep in adolescents. Sleep. 2013 Jun 1;36(6):827-34. doi: 10.5665/sleep.2704. PMID 23729925
- [Background] Taheri S. The link between short sleep duration and obesity: we should recommend more sleep to prevent obesity. Arch Dis Child. 2006 Nov;91(11):881-4. doi: 10.1136/adc.2005.093013. PMID 17056861
- [Background] Rendall MS, Weden MM, Fernandes M, Vaynman I. Hispanic and black US children's paths to high adolescent obesity prevalence. Pediatr Obes. 2012 Dec;7(6):423-35. doi: 10.1111/j.2047-6310.2012.00080.x. Epub 2012 Aug 21. PMID 22911935
- [Background] Singh GK, Kogan MD, Yu SM. Disparities in obesity and overweight prevalence among US immigrant children and adolescents by generational status. J Community Health. 2009 Aug;34(4):271-81. doi: 10.1007/s10900-009-9148-6. PMID 19333745
- [Background] Martinez SM, Thompson-Lastad A. Latino Parents' Insight on Optimal Sleep for Their Preschool-Age Child: Does Context Matter? Acad Pediatr. 2015 Nov-Dec;15(6):636-43. doi: 10.1016/j.acap.2015.07.003. Epub 2015 Sep 26. PMID 26547544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on June 17, 2018 and ended March 9, 2020. Participants were recruited from local San Francisco nonprofit organizations, after school programs, local community events, a federally-qualified community health center and UCSF health clinics.
Groups:
- Short Sleep: This condition required sleeping for less than 8 hours per night for one week.
- Long Sleep: This condition required sleeping for more than 10 hours per night for one week.
Period: Overall Study
Arm/Group | Short Sleep | Long Sleep
Started | 17 | 17
Completed | 16 | 14
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Sleep | Long Sleep | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 14 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.69 (1.09) | 9.74 (.70) | 9.71 (.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 30
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — San Francisco Bay Area participants based on eligibility requirement
  participants
    United States | 16 | 14 | 30
BMI z-score [Mean (Standard Deviation); unit: BMI z-score: 0 is the population average] — BMI z-score of 0 represents the population mean. Clinical cut-offs for overweight risk: BMI z-score greater than +1.0; overweight: BMI z-score greater than +2.0; obese: BMI z-score greater than +3.0.
  BMI z-score: 0 is the population average | 1.57 (1.28) | 2.17 (1.21) | 1.83 (1.26)
Sleep duration [Mean (Standard Deviation); unit: hours per night] — Sleep duration was assessed by maternal report of child's usual time to bed and time to wake up.
  hours per night | 9.69 (.73) | 10.32 (1.68) | 9.99 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Differences in Sleep Duration by Sleep Condition.
Description: Sleep duration will be measured with accelerometers.
Time Frame: One week
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Short Sleep | Long Sleep
Number analyzed (Participants) | 16 | 14
hours | 8.4 (.8) | 8.9 (.6)

2. Primary Outcome: Differences in Physical Activity (Outcome) by Short and Long Sleep Condition.
Description: Physical activity will be measured with accelerometers. Accelerometer data will be used to calculate moderate- to vigorous-intensity physical activity (MVPA; minutes). Activity counts were summed for each 24-hour period categorized into moderate to vigorous levels of physical activity according to the previously established thresholds. Moderate physical activity was set at 0.04 < AEE < 0.10 kcal.kg-1.min-1 or 3.0 < PAR < 6.0, reflective of medium exertion in the standing position. Vigorous physical activity was set at AEE > 0.10 kcal.kg-1.min-1 or PAR > 6.0, reflective of activities at a high level of exertion in the standing position. Moderate-intensity and vigorous-intensity physical activity were combined and expressed as minutes spent in MVPA.
Time Frame: One week
Population: minutes of daily moderate to vigorous physical activity
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Short Sleep | Long Sleep
Number analyzed (Participants) | 16 | 14
minutes | 27 (20) | 30 (17)

3. Primary Outcome: Differences in Carbohydrate Intake by Long and Short Sleep Condition.
Description: Sleep duration will be measured with accelerometers. Eating/dietary intake (outcome) will be assessed on Thursdays and Fridays using 24-hour recalls using Nutrition Data System for Research. Sleep duration will be measured with accelerometers. Dietary intake (outcome) will be assessed on Thursdays and Fridays using 24-hour recalls using Nutrition Data System for Research. Daily sugar intake (grams) will be calculated.
Time Frame: One week
Population: average carbohydrate intake
Measure: Mean (Standard Deviation); unit: kcals
Arm/Group | Short Sleep | Long Sleep
Number analyzed (Participants) | 16 | 14
kcals | 1312 (484) | 1526 (871)

4. Primary Outcome: Differences in Added Sugar Intake by Long and Short Sleep Condition.
Description: as for outcome 3
Time Frame: One week
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Short Sleep | Long Sleep
Number analyzed (Participants) | 16 | 14
grams | 62 (38) | 65 (55)

5. Secondary Outcome: Maternal Sleep Duration
Description: Mothers' bedtimes and wakeup times will be assessed by self report.
Time Frame: Baseline measurement (one time point)
Population: Mothers' reported sleep.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Short Sleep | Long Sleep
Number analyzed (Participants) | 16 | 14
hours | 5.91 (2.15) | 7.56 (3.53)

6. Secondary Outcome: Sleep Hygiene Related to Children's Sleep Schedules.
Description: Sleep hygiene will be assessed by whether the child shares a bed, shares a room and a bed, shares a room (but not a bed), or does not any. Child sleep schedule (bedtime) will be measured by parent report.
Time Frame: Baseline measurement (one time point)
Population: Number of participants who watched TV in bed as a nighttime routine at least once per week.
Measure: Count of Participants; unit: Participants
Arm/Group | Short Sleep | Long Sleep
Number analyzed (Participants) | 16 | 14
Participants | 7 | 9

ADVERSE EVENTS:
Time Frame: No adverse events occurred during the duration of the study (1 year, 9 months).
Arm/Group | Short Sleep | Long Sleep
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT03947918/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03947918/SAP_001.pdf
  • Informed Consent Form (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT03947918/ICF_002.pdf